CLINICAL TRIAL: NCT06027424
Title: The Changes in Blood Pressure in Patients With Obstructive Sleep Apnea Following an Overnight Sleep
Brief Title: Blood Pressure and Obstructive Sleep Apnea
Status: Completed | Type: Observational
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022-07-013CC
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: The Effects of Obstructive Sleep Apnea on Blood Pressure Measurement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Non-OSA: AHI < 5 events/h (AHI, apnea-hypopnea index, the number of apneas and hypopneas per hour of total sleep time)
- Mild OSA: 5 events/h ≤ AHI < 15 events/h
- Moderate OSA: 15 events/h ≤ AHI < 30 events/h
- Severe OSA: AHI ≥ 30 events/h

INTERVENTIONS:
Other:  — observational study, no intervention

SUMMARY:
Bidirectional and causal relationship exists between obstructive sleep apnea (OSA) and hypertension in a dose-response manner, independent of confounding variables such as age, smoking, and body mass index. OSA is conventionally diagnosed and graded by apnea-hypopnea index (AHI). The relationship between AHI and changes of blood pressure deserves further investigation.

DETAILED DESCRIPTION:
Approximately 50% of patients with obstructive sleep apnea (OSA) have hypertension; up to 30% of patients with hypertension have OSA, and the prevalence is even higher in those of resistant hypertension. OSA is conventionally diagnosed and graded by apnea-hypopnea index (AHI). This retrospective study aimed to determine if OSA severity and AHI have effect on blood pressure measurements and the nocturnal changes following an overnight sleep.

ELIGIBILITY:
Inclusion Criteria:

(1). Individuals who underwent full-night polysomnography at Taipei VGH for symptoms related to obstructive sleep apnea, such as snoring and daytime somnolence; (2). Feasibility to measure BP via wrist monitors; (3). Confirmation of wakefulness through electroencephalography.

Exclusion Criteria:

(1). Failure to measure BP via wrist monitors; (2). Age younger than 18 years; (3). Sleep efficiency less than 50%; (4). Central sleep apnea ≥ 50%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who underwent full-night polysomnography at Taipei VGH for symptoms related to obstructive sleep apnea, such as snoring and daytime somnolence
Sampling Method: Non-Probability Sample
Enrollment: 2037 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-07-16 (Actual)

PRIMARY OUTCOMES:
Blood pressure, before sleep and after awakening | 20:30 pm ~ 06:00 am next day
  Measurement of blood pressure at two time points: before sleep and after awakening

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No